CLINICAL TRIAL: NCT03580278
Title: A Safety, Tolerability, Pharmacokinetic, and Efficacy Study of ABY-035/AFO2 Given as Multiple Doses in Sequential Escalating Dose Cohorts in Psoriasis Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetic, and Efficacy of ABY-035/AFO2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Affibody (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABY-035-101
Record Dates: First submitted 2018-05-31; First posted 2018-07-09 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2020-11

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: An exploratory, clinical study with 2 open-dose cohorts is designed to analyze the safety, tolerability, PK, and efficacy of ABY-035/AFO2 in the treatment of subjects with active plaque psoriasis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1:75 mg ABY-035/AFO2 (Experimental): Cohort 1: 75 mg ABY-035/AFO2, once daily for 14 days
  Interventions: Biological: ABY-035/AFO2
- Cohort 2: 150 mg ABY-035/AFO2 (Experimental): Cohort 2: 150 mg ABY-035/AFO2 once daily for up to 28 days
  Interventions: Biological: ABY-035/AFO2

INTERVENTIONS:
Biological: ABY-035/AFO2 — Analyze the safety, tolerability, PK, and efficacy of ABY-035/AFO2 that 25 subjects will receive for treatment of their active plaque psoriasis

SUMMARY:
The purpose of this first-in-human study of the formulation ABY-035/AFO2 is to investigate the safety, tolerability and efficacy after multiple doses in sequential escalating dose cohorts in psoriasis subjects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with plaque psoriasis at least 6 months prior to Screening, if suitable for systemic treatment or phototherapy, and if have a stable active plaque-type psoriasis (stable is defined as without clinically significant flares during the 12 weeks before the first dose). Subjects with psoriatic arthritis may be included if they have not received systemic treatment within the last 12 months and their disease is stable
* Subjects must use adequate contraceptive measures from the Screening Visit until 4 weeks after final administration of the investigational product
* Subject that has a maximum body weight of 243 pounds (110 kg)

Exclusion Criteria:

* Subjects with psoriatic arthritis that have received systemic treatment within the last 12 months.
* Subjects will not be eligible if they have current forms of psoriasis other than chronic plaque-type (e.g. erythrodermic, guttate, or pustular)
* Subject that has a current drug-induced psoriasis form (e.g. a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium)
* Subject that has a history of recurrent or medically important infections, a clinically significant candida infection or clinically significant skin infection with Staphylococcus aureus requiring systemic treatment in the last 12 months prior to the first administration of study drug
* Subject that smokes more than 15 cigarettes, or equivalent in tobacco, per day Subject with a history of suicide attempt or suicidal behavior
* Any live vaccination within 3 months prior to Screening
* Subject that is pregnant, intends to become pregnant during the course of the study, or is lactating

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment-related Adverse Events as assessed by the principles of Common Terminology Criteria for Adverse Events (CTCAE) | 28 Days
  5 male and female psoriasis subjects will be enrolled to obtain who complete treatment or drop out due to adverse events for Cohorts 1 and 2
Number of subjects with treatment-related Adverse Events as assessed by the principles of Common Terminology Criteria for Adverse Events (CTCAE) | 42 Days
  20 male and female psoriasis subjects will be enrolled to obtain who complete treatment or drop out due to adverse events for Cohort 3

SECONDARY OUTCOMES:
Subjects´ level of anti-drug antibodies (ADAs) in the blood | 14 Days dosing period for Cohort 1, 28 Days dosing period for Cohort 3 and 14 Days follow-up period for all Cohorts
  To assess the immunogenicity of ABY-035 after multiple doses of ABY 035/AFO2 in psoriasis subjects
If subjects have assessable pharmacokinetics (PK) of ABY-035 | 14 Days dosing period for Cohort 1, 28 Days dosing period for Cohort 3 and 14 Days follow-up period for all Cohorts
  To investigate the peak plasma concentration (Cmax ) of ABY-035 after multiple doses of ABY-035/AFO2 in psoriasis subjects
If subjects have assessable pharmacokinetics (PK) of ABY-035 | 14 Days dosing period for Cohort 1, 28 Days dosing period for Cohort 3 and 14 Days follow-up period for all Cohorts
  To investigate the Area under the curve (AUC) versus time curve of ABY-035/AFO2 in psoriasis subjects
Efficacy assessment: The change of the subjects´ scaling of a selected target plaque from baseline to the last visit | 14 Days dosing period for Cohort 1, 28 Days dosing period for Cohort 3 and 14 Days follow-up period for all Cohorts
  The results will be summarized as number and percent by visit. Tables from baseline will be prepared for all timepoints
Efficacy assessment: The change of the subjects´erythema of a selected target plaque from baseline to the last visit | 14 Days dosing period for Cohort 1, 28 Days dosing period for Cohort 3 and 14 Days follow-up period for all Cohorts
  The results will be summarized as number and percent by visit. Tables from baseline will be prepared for all timepoints
Efficacy assessment: The change of the subjects´ thickness of a selected target plaque from baseline to the last visit | 14 Days dosing period for Cohort 1, 28 Days dosing period for Cohort 3 and 14 Days follow-up period for all Cohorts
  The results will be summarized as number and percent by visit. Tables from baseline will be prepared for all timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Tooraj Raoof, MD, Principal Investigator — Encino Research Center
Locations (1):
- Raoof, Joseph, Encino, California, United States

IPD SHARING:
Plan to Share IPD: No